CLINICAL TRIAL: NCT01527578
Title: Functional Common Acquisition Protocol Phase of the Simons VIP
Brief Title: Simons Variation in Individuals Project, Functional Common Acquisition Protocol
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: Simons VIP F-CAP
Record Dates: First submitted 2012-01-31; First posted 2012-02-07 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Healthy children; Healthy adults; individuals ages 7-60

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The University of California, San Francisco (UCSF) Simons Variation in Individuals Project (Simons VIP) is currently recruiting healthy controls for a study aimed at better understanding autism spectrum disorder. The UCSF site of the Simons VIP is conducting functional and structural imaging, neuropsychological evaluation, genetic testing, and neurologic exams in healthy individuals to compare with findings in autism spectrum disorder.

DETAILED DESCRIPTION:
To better understand autism spectrum disorders, the UCSF Simons VIP team is recruiting healthy controls to participate in a study involving brain imaging and psychological assessments and questionnaires. The study will involve phone interviews, cognitive testing and questionnaires, genetic testing, physical exam, photographs, non-invasive brain imaging sessions (MRI and MEG). The study can take up to 17 hours to complete, and there may be up to 5 study visits to UCSF and UC Berkeley.

ELIGIBILITY:
Inclusion Criteria:

* Healthy persons age 7 and older
* Must use English as primary language
* Must be able to lie still in MRI scanner for two hours
* Must be willing to travel to UCSF and UC Berkeley for up to 5 study visits.

Exclusion Criteria:

* Any metal implanted in the body
* Extensive dental work
* History of psychiatric of neurological illness
* History of drug or alcohol abuse

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy individuals ages 7 through 60.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Sherr, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States